CLINICAL TRIAL: NCT05724641
Title: Arterial Spin Labeling MRI for Assessing Blood Perfusion in the Human Eye Repeatability Study and Clinical Application
Acronym: PerfRet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CUSL-2022-PerfRet; 2022/06DEC/471 (Other: CEHF)
Record Dates: First submitted 2022-12-15; First posted 2023-02-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Retinal Diseases
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Volunteers (Experimental): N = 10, who do not use contact lenses or eye glasses and have a recent evaluation of vision 10/10 ta participate in the repeatability study.
  Interventions: Diagnostic Test: MRI perfusion imaging using ASL's non-invasive technique
- Chronic (Experimental): N = 30 (10 patients with thyroid associated orbitopathy (TAO), 10 patients with inflammatory optic neuropathy (ION), 10 patients with ischemic neuropathy), all chronic patients followed in ophthalmology consultation, enlightened volunteers ta participate in the study, and presenting a decrease in residual visual acuity entering the TAO, inflammatory or ischemic frameworks.
  Interventions: Diagnostic Test: MRI perfusion imaging using ASL's non-invasive technique
- Acute (Experimental): N = 30 (10 patients with TAO, 10 patients with ION, 10 patients with ischemic neuropathy) all patients seen in the acute phase in ophthalmology consultation who will accept participation in the study, knowing the constraint of repeating the examination in the chronic phase.
  Interventions: Diagnostic Test: MRI perfusion imaging using ASL's non-invasive technique

INTERVENTIONS:
Diagnostic Test: MRI perfusion imaging using ASL's non-invasive technique — Patients will undergo through an MRI-scan using the ASL MRI sequence, as described per protocol.

SUMMARY:
The MRI perfusion imaging using arterial spin labeling (ASL)'s non-invasive technique (i.e. without injection of contrast medium) allows, thanks to recent technological improvement of the spatial resolution, measuring several perfusion parameter of the retinal tissue such as the regional Blood Flow (rBF) or the cerebral blood flow (cBF) expressed in ml/100g/min. Reliable application of ASL thus requires the precision and specificity of the MRI protocol to be tested.

ELIGIBILITY:
Inclusion criteria:

* Carrier of target pathologies: TAO optic neuropathy, inflammatory optic neuropathy, ischemic optic neuropathy.
* no cardiovascular risk factors or other ophthalmological pathology
* adhere to the study protocol after reading the patient information document
* signe the informed consent form to participate in the study
* do not have any contraindications to an MRI examination

Exclusion criteria

* Usual contraindications to MRI (Pacemaker, Metallic foreign body, Cochlear implant,…)
* Severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Repeatability measurement on volunteers | 2 month
  implementing a protocol based on 2 imaging sessions : 1st session with 2 ASL sequences and a 2nd session scheduled 5-7 days later in similar conditions including 1 ASL in volunteers will be applied. This protocol allows assessing the intra-day and the inter-day variability of the measurements using Intra-Class Correlation Coefficient and metric derived from Bland-Altman plots. A total of 20 MRI examinations are planned for this phase of the study.

SECONDARY OUTCOMES:
Mesurement of the retinal perfusion by MRI ASL in patient in acute phase | 4 years
  Analysing the retinal perfusion by ASL to be able to figure out if the decreased visual acuity has an ischemic etiology.
Mesurement of the retinal perfusion by MRI ASLin patient in a chronic phase | 4 years
  Following up the disease process (stability, progression or reversal of the decrease in visual acuity).

CONTACTS AND LOCATIONS:
Overall Officials: Idil Günes-Tatar, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No